CLINICAL TRIAL: NCT03844256
Title: A Phase 1b-2 Study of Mitomycin-c/ Capecitabine ChemoRadiotherapy Combined With Nivolumab Monotherapy or Ipilumimab and Nivolumab, as Bladder Sparing Curative Treatment for Muscle Invasive Bladder Cancer: the CRIMI Study
Brief Title: A Study of Mitomycin-c/ Capecitabine ChemoRadiotherapy Combined With Nivolumab Monotherapy or Ipilumimab and Nivolumab, as Bladder Sparing Curative Treatment for Muscle Invasive Bladder Cancer: the CRIMI Study
Acronym: CRIMI
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Adriaan D. Bins, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CA2099TT
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Urinary Bladder Cancer; Invasive Bladder Cancer
Keywords: Immunotherapy; Chemoradiotherapy; Nivolumab; Ipilimumab; bladder sparing treatment
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Nivolumab; Mitomycin; Capecitabine; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Patients will be treated with radiation therapy over 4 weeks and receive MMC IV on day1 of radiation therapy and capecitabine on each day of radiation therapy as radiosensitizers.
  Phase-1b: enrollment of maximum of 30 patients with a maximum of 10 patients per treatment regimen, in order to determine optimal regimen based on the occurrence of dose limiting toxicities (DLT).
  * Regimen-A: immunotherapy (w1-12) consists of nivolumab 480mg (fixed dose), on day(d)1, d29 and d57.
  * Regimen-B: immunotherapy (w1-12) consists of ipilimumab 1 mg/kg together with Nivolumab 3mg/kg on d1, d22, d43 and d65.
  * Regimen-C: immunotherapy (w1-12) consists of ipilimumab 3 mg/kg and nivolumab 1 mg/kg on d1, d22, d43 and d65.
  All study participants can opt for an additional 10 administrations of nivolumab 480mg fixed dose at intervals of 4 weeks, from week 13 to week 52.
  Phase-2: enrollment of an additional 20 subjects at the regimen determined to be optimal in the phase-1b part.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regimen A (Experimental): Nivolumab monotherapy at 480mg fixed dose administered intravenously (IV) over 60 minutes every 4 weeks for 3 doses.
  All study participants can opt for an additional 10 administrations of nivolumab 480mg fixed dose at intervals of 4 weeks, from week 13 to week 52.
  Interventions: Combination Product: nivolumab 480mg
- Regimen B (Experimental): Nivolumab at 3 mg/kg administered IV over 60 minutes combined with ipilimumab at 1 mg/kg administered IV over 90 minutes every 3 weeks for 4 doses.
  All study participants can opt for an additional 10 administrations of nivolumab 480mg fixed dose at intervals of 4 weeks, from week 13 to week 52.
  Interventions: Combination Product: nivolumab 3mg/kg, ipilimumab 1mg/kg
- Regimen C (Experimental): Nivolumab at 1 mg/kg administered IV over 60 minutes combined with ipilimumab at 3 mg/kg administered IV over 90 minutes every 3 weeks for 4 doses.
  All study participants can opt for an additional 10 administrations of nivolumab 480mg fixed dose at intervals of 4 weeks, from week 13 to week 52.
  Interventions: Combination Product: nivolumab 1mg/kg, ipilimumab 3mg/kg

INTERVENTIONS:
Combination Product: nivolumab 480mg — Immuno-chemoradiotherapy
  Other Names: mitomycin-c 12mg/m2 IV; capecitabine 750mg/m2; radiotherapy 40Gy in 20 fractions of 2Gy
  Arms: Regimen A
Combination Product: nivolumab 3mg/kg, ipilimumab 1mg/kg — Immuno-chemoradiotherapy
  Other Names: mitomycin-c 12mg/m2 IV; capecitabine 750mg/m2; radiotherapy 40Gy in 20 fractions of 2Gy
  Arms: Regimen B
Combination Product: nivolumab 1mg/kg, ipilimumab 3mg/kg — Immuno-chemoradiotherapy
  Other Names: mitomycin-c 12mg/m2 IV; capecitabine 750mg/m2; radiotherapy 40Gy in 20 fractions of 2Gy
  Arms: Regimen C

SUMMARY:
A multicenter Phase 1b/2, two stage, open label study of MMC/Capecitabine ChRT combined with nivolumab monotherapy or nivolumab and ipilimumab combination therapy in adult (>18 years) subjects with non-metastatic muscle invasive bladder cancer that qualify for ChRT with curative intent.

DETAILED DESCRIPTION:
Immunotherapy combined with chemoradiation for localized bladder cancer may exhibit improved efficacy with an acceptable toxicity profile.

The aim of this phase 1b/2, two stage, open label study of MMC/Capecitabine ChRT combined with nivolumab monotherapy or nivolumab and ipilimumab combination therapy stuy is: to assess the feasibility and safety, the disease free survival (DFS) and disease free survival rate (DFS-rate) of the addition of nivolumab and/or ipilimumab to MMC/capecitabine chemoradiation of the bladder.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Wish to preserve their bladder function or be ineligible for cystectomy.
* Must have undergone transurethral biopsy of the bladder tumor, within 35 days of planned treatment commencement. The patient should have a histologically-confirmed diagnosis of muscle-invasive T2-T4a, N0-1M0 urothelial cell carcinoma of the bladder.
* Must have undergone maximal transurethral resection of the bladder tumour, to an extent that is judged as safe by the urologist performing the resection, within 35 days of planned treatment commencement.
* Subjects with tumors of mixed urothelial/non-urothelial cell histology are allowed, but urothelial cell carcinoma must be the predominant histology (>50%). Subjects with predominant or exclusively non-urothelial cell histology are not allowed.
* Have planned for chemoradiotherapy as definitive treatment.
* Have a performance status of 0 or 1 on the ECOG Performance Scale
* Have a bladder function that is accessible for cystoscopical follow up.
* Demonstrate adequate organ function. All screening labs should be performed within 28 days of registering the patient on the trial.
* Female participants of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to registering the patient. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female participants of childbearing potential should be willing to one highly effective method of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 5 month after the last dose of study medication Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male participants should agree to use condoms starting with the first dose of study therapy through 7 month after the last dose of study therapy.
* Willing to consent to the use of their collected tumor specimen, blood and urine as detailed in the protocol for future scientific research including but not limited to DNA, RNA and protein based biomarker detection.

Exclusion Criteria:

* Has DPD deficiency.
* Has concurrent extra-vesical (i.e. urethra, ureter or renal pelvis) urothelial cell carcinoma of the urothelium. Patients who have involvement of the prostatic urethra with urothelial cell cancer may be included if the location can be safely incorporated in the radiation field.
* Extensive or multifocal bladder carcinoma in situ (CIS) precluding curative chemoradiotherapy.
* Evidence of distant metastatic disease on a CT or FDG PET/CT chest/abdomen/pelvis performed within 28 days prior to study entry. Up to 3 metastatic lymphnodes in the pelvis (below the common iliac arteries) are allowed, if these can be incorporated in the radiotherapy field.
* Prior pelvic lymph-adenectomy
* Prior pelvic radiotherapy
* Has had prior intravenous chemotherapy, targeted small molecule therapy, or radiation therapy for treatment of bladder cancer. Prior intravesical use of BCG and MMC is permissible.
* Unsuitable for concurrent MMC / capecitabine based ChRT based on pre-existing medical conditions.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy over 10mg daily prednisone (or equivalent) or any other form of immunosuppressive therapy within 14 days prior to registering the patient. Patients with adrenal insufficiency receiving replacement dose steroids are allowed on the trial.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to nivolumab and/or ipilimumab or any of its excipients.
* Prior or concurrent known additional malignancy of any site unless disease free for 5 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, Stage T1a well differentiated prostatic carcinoma in men (Gleason = 3+3, PSA <5)
* Has any history of active autoimmune disease, Stevens-Johnson syndrome or Guillain-Barre. Exceptions to this are:

  1. Patients with autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone
  2. Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has an Human Immunodeficiency Virus (HIV) infection with a PCR detectable viral load.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Toxicity scored with CTCAE v 4.03 | 6 weeks after start of the combination therapy
  Toxicity scored with CTCAE v 4.03
Incidence of dose limiting toxicity (DLT) | 6 weeks after start of combination therapy
Disease free survival (DFS) | 5 years
disease free survival-rate (DFS-rate) | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Overall survival rate | 5 years
Response rate | up to 5 years
  Cystoscopy at week 12 and week 24 will be performed. From week 12 onward 3-montly CT scans will be done in the context of the current standard of care up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan D. Bins, MD PhD, Principal Investigator — Amsterdam UMC, AMC
Locations (3):
- Netherlands (3):
  - Amsterdam UMC, VUmc, Amsterdam, North Holland
  - Amsterdam UMC, AMC, Amsterdam, North Holland
  - LUMC, Leiden, South Holland

IPD SHARING:
Plan to Share IPD: No